CLINICAL TRIAL: NCT01344408
Title: Effectiveness of Computer Assisted Training in Vestibular Rehabilitation for Older Patients With Vestibular Dysfunction
Brief Title: Effectiveness of Computer Assisted Training for Older People With Vestibular Dysfunction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M-20090189
Record Dates: First submitted 2010-03-15; First posted 2011-04-29 (Estimated); Last update posted 2016-05-20 (Estimated); Status verified 2015-10

CONDITIONS: Dysfunction of Vestibular System
Keywords: Dizziness; rehabilitation; geriatric; IT-technology
MeSH Terms: conditions — Dizziness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Computer-training (Experimental): The computer-training program, Move it to improve it was installed in the participants homes using an internet-connected computer with a web camera connected to a cloud-based specifically adapted interactive training program.
  Interventions: Procedure: Computer-training
- Printed instructions (Experimental): A training program delivered as printed instructions
  Interventions: Procedure: Computer-training

INTERVENTIONS:
Procedure: Computer-training — The computer-training program "Move IT To Improve IT" is a exercise program which is installed and used on a Apple Imac in the patients home to support vestibular rehabilitation
  Other Names: Move It To Improve IT

SUMMARY:
BACKGROUND A Cochrane review from 2003 found that about 30% of people 65 years or older each year fall and that number is even higher for elder people living in institutions. Falls are the cause of 95% of all hip fractures, resulting in prolonged hospitalization and prolonged disability. In patients who are referred to the emergency room after unexplained fall, a study of 564 patients showed that 80% of the patients had vestibular symptoms characterized by balance problems, nausea, impairment, vomiting, and dizziness. 41% of the patients had dizziness suggesting a dysfunctional vestibular system called vestibular dysfunction. In patients with vestibular dysfunction, vestibular rehabilitation (VR) can reduce fall risk. Several studies show however that the elderly has a decreased compliance in relation to the performance of home exercise.

A solution to support the older vestibular rehabilitation process and to maintain the achieved level of functionality after the rehabilitation process is the computer-training program "Move It To Improve It" (MITII). Based on individual studies and tests therapists develop a personalized rehabilitation program permanently corrected, modified and adjusted. The system generates feedback to the therapists at hospital with information about the person's daily training and scores of individual exercises. The Web cam makes it possible to make video footage and pictures to be used in the feedback information. The system also establish direct communication between users and therapists. The web community provide the framework for a telerehabilitation system, which means that the hospital can service more users in the same period.

The ph.d. consist of three studies which has the purposes:

To compare a computer exercise program (Mitii) with conservative home-training according to printed instructions in the rehabilitation of patients with vistibular dysfunction in an outpatient clinic To investigate whether the effect of vestibular rehabilitation is preserved three months after the completion of supervised training in an outpatient clinic for specific vestibular rehabilitation and whether a computer assisted home training program (Mitii) is superior to printed instructions in this respect To evaluate patient experience and barriers for the use fo the computer assisted rehabilitation of patients with vestibular dysfunction

DETAILED DESCRIPTION:
BACKGROUND A Cochrane review from 2003 found that about 30% of people 65 years or older each year fall and that number is even higher for elder people living in institutions. Falls are the cause of 95% of all hip fractures, resulting in prolonged hospitalization and prolonged disability. Half of the elderly who incurs hip fracture will never be able to walk like they did before the fall, and one year mortality is between 15 and 25%. Meanwhile, the population 65 years old and older are increasing and the National Institute of Aging notes in a 2001 report that the world's population of 65 years old and older is growing by 800.000 a year. It is estimated that the cost of fall-related accidents in 2020 will reach $54.9 billion in the U.S. alone.

In patients who are referred to the emergency room after unexplained fall, a study of 564 patients showed that 80% of the patients had vestibular symptoms characterized by balance problems, nausea, impairment, vomiting, and dizziness. 41% of the patients had dizziness suggesting a dysfunctional vestibular system called vestibular dysfunction. A study in 6785 participants included the National Health and Nutrition Examination Surveys in the U.S. showed that the prevalence of vestibular dysfunction increases significantly with age. The prevalence for vestibular dysfunction among participants aged 60-69 years was 49.4%, 68,7% among participants aged 70-79 and 84,8% for the participants aged 80 years or older.

In patients with vestibular dysfunction, vestibular rehabilitation (VR) can reduce fall risk. In 2007 a large Cochrane review compared randomized studies of VR, where the authors concluded that there is moderate to strong evidence of the efficacy of VR. Several authors describe that the reduction of the patient's dizziness in VR only can be achieved by simultaneous establishment of daily exercises at home. Several studies show however that the elderly has a decreased compliance in relation to the performance of home exercise.

A solution to support the older vestibular rehabilitation process and to maintain the achieved level of functionality after the rehabilitation process is the computer-training program "Move It To Improve It" (MITII). The program has been successfully used for home training of patients with cerebral palsy and is composed of exercises that are both motivating and guiding.

Based on individual studies and tests therapists developed a personalized rehabilitation program permanently corrected, modified and adjusted for vestibular dysfunction patients. The system could generate feedback to the therapists at hospital with information about the person's daily training time. Basic element in MITII is an exercise. As an example the exercise could be to catch an insect with a net using head movements. Management method is drag-and-drop, which means that management of the network is done by the user with a colour which can retain and move objects on the screen.

PURPOSE

The study consist of three studies which has the purposes:

To compare a computer exercise program (Mitii) with conservative home-training according to printed instructions in the rehabilitation of patients with vistibular dysfunction in an outpatient clinic To investigate whether the effect of vestibular rehabilitation is preserved three months after the completion of supervised training in an outpatient clinic for specific vestibular rehabilitation and whether a computer assisted home training program (Mitii) is superior to printed instructions in this respect To evaluate patient experience and barriers for the use fo the computer assisted rehabilitation of patients with vestibular dysfunction

METHODS

The study consists of three parts:

1. A randomized study where the aim is to examine whether Mitii can improve the outcome of vestibular rehabilitation.The study includes 31 patients in a control and 32 patients in a intervention group with vestibular dysfunction. The control group undergoing normal rehabilitation in the fall clinic (ie, 2 times weekly rehabilitation in the fall clinic + home exercise program with printed instructions) while the intervention group undergoes rehabilitation with MITII (ie 2 times weekly rehabilitation in the fall clinic + MITII to support home exercises. The expectation is that the intervention group improve the most.
2. After completion of the rehabilitation period the patients must maintain their functionality by home exercises. The patients in the intervention group keeps MITII in further 12 weeks to compare with control group of patients who have had a traditional exercise program as printed instructions available. The expectation is that the intervention group will be able to maintain their functionality best.
3. The last part of the study will be qualitative to study how the elderly feel about using IT support in their own homes. This qualitative study will consist of interviews of 7 patients included in the intervention group.

STUDY POPULATION Patients referred to the fall clinic from their GP or Casualty department, Aarhus University Hospital. A geriatric doctor will examine and evaluate what underlies the patient's fall issue. The patients who are diagnosed by vestibular dysfunction and are accepting to take part of the project, refers to the Ear, nose and throat department H, Aarhus University Hospital for verification of the vestibular dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Patient Acceptance
* 65 years old or older
* Peripheral vestibular dysfunction, stable (ie no inflammatory processes ie neuronitis vestibulitis and/or fluctuations symptoms ie Meniere)
* Central vestibular dysfunction without other co-morbidities (eg. Parkinson's, Stroke)
* Mixed peripheral and central vestibular dysfunction without other co-morbidity

Exclusion Criteria:

* Lack of vision
* If exercise therapy is contraindicated
* Significant cardiac problems
* Taking medicine with risk of vestibular side effects (benzodiazepines, sedatives)
* Dementia (MMSE test <27 or an anamnesis suggesting dementia)
* Stroke within the past 6 months
* Other cognitive dysfunction
* Operation of hip fractures within the last 3 months

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2010-01; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Static balance will be measured by the "One leg Stand test" | 16 weeks of rehabilitation
  Static balance

SECONDARY OUTCOMES:
Dynamic balance will be measured by the "Dynamic Gait Index" | 8, 16 and 28 weeks of rehabilitation
  Dynamic balance
Experienced dizziness handicap will be measured by the "Dizziness Handicap Inventory" | 8, 16 and 28 weeks of rehabilitation
  Experienced dizziness handicap
Static balance will be measured by the "Modified Clinical Test of Sensory Interaction and Balance". | 8, 16 and 28 weeks of rehabilitation
  Static balance
Quality of life will be measured by the "SF-12" | 8, 16 and 28 weeks of rehabilitation
  Quality of life
Under extremities strength test will be measured by the "Chair Stand Test" | 8, 16 and 28 weeks of rehabilitation
  Under extremities strength testing
Motion triggered dizziness will be measured by the "Motion Sensitivity Test" | 8, 16 and 28 weeks of rehabilitation
  Motion triggered dizziness
Dizziness will be measured by the "Visual Analogue Scale" | 8, 16 and 28 weeks of rehabilitation
  Dizziness scores on the Visual Analogue Scale

CONTACTS AND LOCATIONS:
Overall Officials: E.M. Damsgaard, Study Chair — Geriatric Section; M. Brandt, Principal Investigator — Geriatric Section
Locations (1):
- Aarhus Hospital, Aarhus, Aarhus C, Denmark

REFERENCES:
- [Background] Gillespie LD, Gillespie WJ, Robertson MC, Lamb SE, Cumming RG, Rowe BH. Interventions for preventing falls in elderly people. Cochrane Database Syst Rev. 2003;(4):CD000340. doi: 10.1002/14651858.CD000340. PMID 14583918
- [Background] Grisso JA, Kelsey JL, Strom BL, Chiu GY, Maislin G, O'Brien LA, Hoffman S, Kaplan F. Risk factors for falls as a cause of hip fracture in women. The Northeast Hip Fracture Study Group. N Engl J Med. 1991 May 9;324(19):1326-31. doi: 10.1056/NEJM199105093241905. PMID 2017229
- [Background] Pothula VB, Chew F, Lesser TH, Sharma AK. Falls and vestibular impairment. Clin Otolaryngol Allied Sci. 2004 Apr;29(2):179-82. doi: 10.1111/j.0307-7772.2004.00785.x. PMID 15113307
- [Background] Agrawal Y, Carey JP, Della Santina CC, Schubert MC, Minor LB. Disorders of balance and vestibular function in US adults: data from the National Health and Nutrition Examination Survey, 2001-2004. Arch Intern Med. 2009 May 25;169(10):938-44. doi: 10.1001/archinternmed.2009.66. PMID 19468085
- [Background] Macias JD, Massingale S, Gerkin RD. Efficacy of vestibular rehabilitation therapy in reducing falls. Otolaryngol Head Neck Surg. 2005 Sep;133(3):323-5. doi: 10.1016/j.otohns.2005.04.024. PMID 16143174
- [Background] Brandt T. Management of vestibular disorders. J Neurol. 2000 Jul;247(7):491-9. doi: 10.1007/s004150070146. PMID 10993488
- [Background] Hillier SL, Hollohan V. Vestibular rehabilitation for unilateral peripheral vestibular dysfunction. Cochrane Database Syst Rev. 2007 Oct 17;(4):CD005397. doi: 10.1002/14651858.CD005397.pub2. PMID 17943853
- [Background] Krebs DE, Gill-Body KM, Parker SW, Ramirez JV, Wernick-Robinson M. Vestibular rehabilitation: useful but not universally so. Otolaryngol Head Neck Surg. 2003 Feb;128(2):240-50. doi: 10.1067/mhn.2003.72. PMID 12601321
- [Background] van der Bij AK, Laurant MG, Wensing M. Effectiveness of physical activity interventions for older adults: a review. Am J Prev Med. 2002 Feb;22(2):120-33. doi: 10.1016/s0749-3797(01)00413-5. PMID 11818183
- [Background] Forkan R, Pumper B, Smyth N, Wirkkala H, Ciol MA, Shumway-Cook A. Exercise adherence following physical therapy intervention in older adults with impaired balance. Phys Ther. 2006 Mar;86(3):401-10. PMID 16506876
- [Background] Whitney SL, Sparto PJ, Hodges LF, Babu SV, Furman JM, Redfern MS. Responses to a virtual reality grocery store in persons with and without vestibular dysfunction. Cyberpsychol Behav. 2006 Apr;9(2):152-6. doi: 10.1089/cpb.2006.9.152. PMID 16640469
- [Background] Pavlou M, Lingeswaran A, Davies RA, Gresty MA, Bronstein AM. Simulator based rehabilitation in refractory dizziness. J Neurol. 2004 Aug;251(8):983-95. doi: 10.1007/s00415-004-0476-2. PMID 15316804
- [Derived] Smaerup M, Laessoe U, Gronvall E, Henriksen JJ, Damsgaard EM. The Use of Computer-Assisted Home Exercises to Preserve Physical Function after a Vestibular Rehabilitation Program: A Randomized Controlled Study. Rehabil Res Pract. 2016;2016:7026317. doi: 10.1155/2016/7026317. Epub 2016 Feb 11. PMID 26981283
- [Derived] Smaerup M, Gronvall E, Larsen SB, Laessoe U, Henriksen JJ, Damsgaard EM. Computer-assisted training as a complement in rehabilitation of patients with chronic vestibular dizziness--a randomized controlled trial. Arch Phys Med Rehabil. 2015 Mar;96(3):395-401. doi: 10.1016/j.apmr.2014.10.005. Epub 2014 Oct 25. PMID 25450134